CLINICAL TRIAL: NCT06565416
Title: Opioid and Pain Treatment in Indigenous Communities (OPTIC) Trial: Implementation of Screening and Brief Intervention
Brief Title: Opioid and Pain Treatment in Indigenous Communities (OPTIC) Trial
Acronym: OPTIC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2303044342; RM1DA055301 (NIH); 2206007094 (Other: University of New Mexico)
Record Dates: First submitted 2024-08-19; First posted 2024-08-22 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Opioid Use Disorder; Opioid Misuse; Chronic Pain
MeSH Terms: conditions — Opioid-Related Disorders; Chronic Pain

STUDY DESIGN:
Intervention Model Description: A provider-level implementation intervention will be administered at each of the three participating sites. The investigators will examine implementation and effectiveness outcomes before, during, and after implementation.
Who Masked: Participant
Masking Description: Given the single group design, it is not feasible to blind investigators or outcomes assessor. Given that the intervention occurs at the site level among providers, patients/clients can be considered blinded given that they are not the direct target of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Pre-Intervention (No Intervention): Baseline prior to any involvement with the project
- Intervention (No Intervention): A workgroup for each clinic meets for approximately 6 months to select the specific goals for the clinic to be targeted during the implementation phase.
- Implementation (Active Comparator): Evidence-based implementation strategies are put into practice for approximately 6 months.
  Interventions: Behavioral: Implementation Strategies
- Sustainment (No Intervention): Measuring the degree to which the clinic maintains the implementation phase goals.

INTERVENTIONS:
Behavioral: Implementation Strategies — Culturally centering screening and brief intervention for chronic pain and opioid misuse/opioid use disorder among American Indian/Alaska Native clients
  Arms: Implementation

SUMMARY:
The present study seeks to examine the implementation process of culturally tailoring screening and brief intervention for both chronic pain and opioid misuse/opioid use disorder in three American Indian and Alaska Native (AI/AN) serving clinics. The investigators also will assess staff perspectives on this implementation as well as a survey to understand clients at these sites who have chronic pain and opioid misuse/opioid use disorder.

DETAILED DESCRIPTION:
Given the health disparities in AI/AN populations and lack of access to quality care for comorbid chronic pain and opioid misuse/OUD, the proposed study seeks to build upon the strong relationships between the research team and the AI/AN communities. There is a dearth of prior research examining chronic pain, opioid misuse/OUD, and other comorbid conditions (mood disorders, anxiety disorders, other SUD) in AI/AN populations. Using CBPR methods, the investigators will work with the OPTIC Collaborative Board to develop a culturally centered implementation intervention to improve screening and brief interventions with AI/AN clients with chronic pain and opioid misuse/OUD (Phase I, Aim 1). Specifically, in collaboration with the community partners and the OPTIC Collaborative Board, the investigators will develop a provider training to increase provider skills and self-efficacy to focus conversations on managing chronic pain (rather than trying to eliminate it) and improving client functioning within cultural frameworks of wellbeing. The goal is to develop, implement, and evaluate culturally centered implementation strategies to increase screening and brief intervention for chronic pain, opioid misuse/OUD in clinics serving AI/AN communities. The investigators will conduct a type III effectiveness-implementation trial over the course of 24 months at each clinical site utilizing EMR data and longitudinal staff surveys to test the implementation outcomes (Phase II, Aim 2) as well as patient surveys to test effectiveness outcomes (Phase II, Aim 3) . The investigators hypothesize that the culturally centered approach will increase rates of screening and brief intervention, and ultimately improve outcomes among AI/AN clients with chronic pain and OUD who receive treatment in primary care. The investigators also will assess staff perspectives on this implementation as well as a survey to understand clients at these sites who have chronic pain and opioid misuse/opioid use disorder for the purpose of identifying areas of treatment needs, and examining the efficacy of a provider-level implementation intervention delivered at the sites from which our participants will be sampled.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide informed consent
* have English comprehension and proficiency
* receiving services at one of our participating study sites
* report current chronic pain and/or opioid misuse/opioid use disorder
* self-identify as American Indian/Alaska Native

Exclusion Criteria:

* if they have a psychiatric, cognitive, or medical condition that interferes with the consenting process

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Number of clients screened for chronic pain and opioid misuse/opioid use disorder | 6 months (or duration of implementation phase)
  Derived from electronic medical records
Number of clients screened for chronic pain and opioid misuse/opioid use disorder | 6 months (or duration of sustainment phase)
  Derived from electronic medical records

CONTACTS AND LOCATIONS:
Overall Officials: Matthew R Pearson, PhD, Principal Investigator — University of New Mexico
Locations (3):
- United States (3):
  - Clinic Site A (blinded pending tribal approval), Arcata, California
  - Clinic Site C (blinded pending tribal approval), Minneapolis, Minnesota
  - Clinic Site B (blinded pending tribal approval), Toppenish, Washington

IPD SHARING:
Plan to Share IPD: No
Each Tribal partner has would need to agree to have their data shared.